CLINICAL TRIAL: NCT07178236
Title: Evaluation of a Novel Portable Mainstream Capnograph MARIE in Adult Postoperative Patients - A Prospective Feasibility Study
Brief Title: Evaluation of a Novel Portable Capnograph (MARIE) in Adult Postoperative Patients
Acronym: NOVOCAP-Postop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malin Jonsson Fagerlund (Other)
Responsible Party: Sponsor-Investigator, Malin Jonsson Fagerlund, Professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NOVOCAP-Postop; CIV-ID 25-06-053097 (Registry Identifier: Swedish Medical Products Agency)
Record Dates: First submitted 2025-09-06; First posted 2025-09-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Surgery; Anesthesia; Postoperative Care; Respiration Rate Detection; Capnography; Monitoring
Keywords: capnography; Postoperative; surgery; anaesthesia; monitoring; respiration; novel equipment
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MARIE (Experimental): Portable capnograph
  Interventions: Device: MARIE

INTERVENTIONS:
Device: MARIE — Portable capnoghraphy

SUMMARY:
Postoperative respiratory complications are common and sometimes hard to detect early. Desaturation is a late sign of reduced minute ventilation, especially if the patient is on supplemental oxygen, and measurement of arterial or endtidal CO2 will rapidly detect a reduction in minute ventilation. Capnography offers a non-invasive and continuous measure of end-tidal expiratory pressure of carbon dioxide (EtCO2). Capnography is not a standard in postoperative care but rather quite rare. In the present study we evaluate a novel portable capnography device, MARIE, in postoperative patients.

1. The primary outcome is to describe the correlation of end-tidal CO₂ (EtCO₂) measurements between MARIETM (Oxlantics Medical) and Philips Intelli Vue X3 Microstream.
2. Secondary outcomes include

   1. Correlation between PaCO₂ and EtCO₂ measured by MARIE and Philips Intelli Vue X3 Microstream, respectively.
   2. Time trajectories of PaCO₂ and EtCO₂ measured using MARIE and Philips Intelli Vue X3 Microstream, respectively
   3. The overall agreement between the EtCO2 measured by MARIE and Philips Intelli Vue X3 Microstream and PaCO2
   4. Respiratory rate measured by MARIE compared to manual counting and Philips Intelli Vue X3.
   5. Comparison of oxygen flow by MARIE and the rotameter.
   6. Comfort as reported by patient.
   7. Usability as reported by nurse.
   8. Reasons for premature termination of MARIE
   9. Registration of technical problems, for example unexpected shut downs and blockage by mucus.

MARIE will be applied immediately after tracheal extubation after surgery. CO2 values from MARIE will be compared to EtCO2 and PaCO2 derived from capnography equipment routinely used in the hospital and blood gas analysis, at set intervals in the postoperative ward. Respiratory rate will be compared to our standard care monitors, ie Philips Intelli Vue X3, alongside manual counting. Rate of oxygen delivery, when applicable, will also be compared to the rotameter.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, ≥18 years of age
2. Elective surgery under general anesthesia
3. Planned for over night postoperative care

Exclusion Criteria:

1. Tracheostomy
2. Nasal obstruction
3. Rhino- or oral surgery
4. Not able to understand study information or signing consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-09-22 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is correlation of end-tidal CO₂ (EtCO₂) measurements between MARIETM (Oxlantics Medical) and Philips Intelli Vue X3 Microstream | From enrolment to discharge from the postoperative unit or maximum 24 hours
  End-tidal CO₂ (EtCO₂) measurements will be measured by MARIE (Oxlantic Medical AB) and Philips Intelli Vue X3 Microstream at several occasions and thereafter correlated

SECONDARY OUTCOMES:
Correlation between PaCO₂ and EtCO₂ measured by MARIE and Philips Intelli Vue X3 Microstream, respectively. | From enrolment in the study until discharge from the postoperative unit or maximum 24 hours
  Measurement of arterial PCO₂ and EtCO₂ measured by MARIE and Philips Intelli Vue X3 Microstream at the same time will be done repeatedly and thereafter correlated
Time trajectories of PaCO₂ and EtCO₂ measured using MARIE and Philips Intelli Vue X3 Microstream, respectively | From enrolment until discharge from the postoperative unit or maximum of 24 hours
  Arterial PCO₂ and EtCO₂ measured using MARIE and Philips Intelli Vue X3 Microstream will be measured repeatedly and thereafter correlated
The overall agreement between the EtCO2 measured by MARIE and Philips Intelli Vue X3 Microstream and PaCO2 | From enrolment until discharge from the postoperative unit or a maximum of 24 hours
  EtCO2 measured by MARIE and Philips Intelli Vue X3 Microstream and PaCO2 will be collected simultaneously and repeatedly and thereafter investigated
Respiratory rate measured by MARIE compared to manual counting and Philips Intelli Vue X3 | From the enrolment in the study and until discharge from the postoperative unit or a maximum of 24 hours
  Respiratory rate measured by MARIE compared to manual counting and Philips Intelli Vue X3 will be measured simultaneously and thereafter compared and correlated
Comparison of oxygen flow by MARIE and the rotameter | From enrolment in the study until discharge from the postoperative unit or a maximum of 24 hours
  Oxygen flow rate by MARIE and the rotameter will be documented repeatedly and simultaneously and thereafter compared and correlated
Comfort as reported by patient as VAS (0-10). | Three times/24 hours from admission to the postoperative unit until discharge from the postoperative unit or maximum 24 hours
  Comfort by the patient will be scored by the patient three times/24 hours on average Visual Analogue Scale from 1-10. 0= Worst comfort, 10= Comfortable
Usability as reported by nurse as VAS (0-10). | From the time of enrolment until discharge from the postoperative unit of maximum 24 hours
  The nurse will score the usability on a Visual Analogue Scale (VAS) from 0-10. 0=Very low usability, 10=very high usability
Reasons for premature termination of MARIE | From the enrolment to the discharge from the postoperative unit or a maximum of 24 hours
  Report of reasons for premature termination

CONTACTS AND LOCATIONS:
Overall Officials: Malin Jonsson Fagerlund, Professor, Principal Investigator — Karolinska University Hospital & Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided